CLINICAL TRIAL: NCT04651946
Title: Cell-free DNA Methylation for the Diagnosis and Monitoring of Epithelial Ovarian Cancer: The Training and Validation Sets in China
Brief Title: Cell-free DNA Methylation for Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EOC-METHY
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Epithelial Ovarian Cancer; DNA Methylation; Benign Ovarian Tumor; Training Set; Validation Set; Cell-free DNA; Liquid Biopsy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: All eligible patients accept DNA methylation testing in serum and in ovarian tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DNA methylation testing — Methylation testing of host DNA, namely, OPCML, FODX3 and CDH13, in the peripheral serum

SUMMARY:
Liquid biopsy is challenging for the diagnosis of epithelial ovarian cancer (EOC). In this study, we performed the methylation testing of host DNA, namely, OPCML, FODX3 and CDH13, in the peripheral serum to discover the diagnostic and supervision roles of DNA methylation in EOC patients. The study compromises two stages.

In the training set, DNA methylation testing is performed in the ovarian tissues from EOC and paired benign ovarian tumor patients. The cut-off values of methylation are produced in this stage. On the meantime, serum DNA methylation testing is also performed to reveal its accordance and accuracy compared with the results of ovarian tissues.

In the validation set, serum DNA methylation testing is performed in unselected ovarian tumor patients with definite cut-off values to validate its accuracy based on known histology of ovarian tumors.

In training and validation sets, serum DNA methylation is also performed after major surgeries for EOC as to illustrate the changes of methylation testing, therefore, reflection the supervision role of DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* With definite histological diagnosis of epithelial ovarian cancer and paired benign ovarian tumor in training set, and with definite histological diagnosis of ovarian tumor in validation set.
* With sufficient fresh peripheral serum and ovarian samples for DNA methylation testing before with or without after major surgeries.
* Aged 18 years or older.
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2022-11-26 (Estimated)

PRIMARY OUTCOMES:
Cut-off values of targeted DNA methylation in epithelial ovarian cancer | Two years
  The cut-off values are achieve by paired epithelial ovarian cancer and benign ovarian tumor patients.

SECONDARY OUTCOMES:
Accuracy of serum DNA methylation in epithelial ovarian cancer | Two years
  The accuracy is supported by sensitivity, specificity, negative predictive value and positive predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China